CLINICAL TRIAL: NCT06775288
Title: Effect of Hypoglycemia Prevention and Awareness Program (HypoPAP) on Patient Outcomes: Randomized Controlled Trial
Brief Title: Hypoglycemia Prevention and Awareness Program
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Merve DerviAYoAYlu (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Sponsor-Investigator, Merve DerviAYoAYlu, Research Assistant, Dokuz Eylul University
Organization: Dokuz Eylul University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: DokuzEU-IHH-MD-01
Record Dates: First submitted 2025-01-04; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Diabetes; Hypocalcemia; Telehealth; Nursing Care; Nursing Education
Keywords: hypoglycemia awareness; , telehealth; hypoglycemia; type 2 diabetes; nursing care
MeSH Terms: conditions — Diabetes Mellitus; Hypocalcemia; Hypoglycemia; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): 3 months Hypoglycemia Prevention and Awareness Program
  Interventions: Other: Hypoglycemia prevention and awareness program (HypoPAP)
- Control Group (No Intervention): 3 months follow-up

INTERVENTIONS:
Other: Hypoglycemia prevention and awareness program (HypoPAP) — Online hypoglycemia prevention and awareness training Supporting the prevention of hypoglycemia with the use of evidence-based diabetes-friendly plates Encouraging physical activity and supporting glycemic control with a pedometer Filling in a weekly problem-solving notebook Conducting weekly online problem-solving meetings Online counseling service when needed
  Arms: Experimental Group

SUMMARY:
The aim of this project is to examine the effects of the Hypoglycemia Prevention and Awareness Program (HypoPAP) on patient outcomes, including metabolic, psychological, social, and economic parameters, in individuals with type 2 diabetes and impaired hypoglycemia awareness.

Through the interventions provided to participants, the study aims to achieve the following improvements:

* Physiological parameters: Enhanced glycemic control, reduced hypoglycemia frequency, improved hypoglycemia awareness, and optimized HbA1c levels.
* Psychological parameters: Reduced fear of hypoglycemia, increased hypoglycemic confidence, and improved attitudes toward hypoglycemia management.
* Social parameters: Decreased social withdrawal due to fear of hypoglycemia, as assessed through relevant items in validated scales.
* Economic parameters: Reduced frequency of hospitalizations and emergency department visits.

Overall, the program seeks to enhance participants' ability to prevent and manage hypoglycemia, thereby improving their overall well-being.

DETAILED DESCRIPTION:
Optimal diabetes management is a delicate balance between treating hyperglycemia and avoiding the risk of sudden hypoglycemia. Hypoglycemia is a common, recurring, feared, and neglected complication among endocrine emergencies in individuals with diabetes. Intensive glycemic control is very important in preventing microvascular and macrovascular complications of diabetes. However, hypoglycemia is a significant obstacle to effective treatment. Individuals with diabetes experience many chronic microvascular and macrovascular complications. The most challenging and frightening complication for individuals with diabetes and their families is hypoglycemia. Diabetics are afraid of experiencing hypoglycemia, and fear of hypoglycemia is a significant obstacle to achieving normoglycemia. Hypoglycemia in individuals with type 2 diabetes often occurs due to errors in self-management. Hypoglycemia limits the physical activities and daily living activities of individuals with diabetes. Hypoglycemia, which negatively affects the physiological and psychological health of individuals with diabetes, also reduces the quality of life of patients and their families. Hypoglycemia is also the most important limitation of diabetes treatment. As the severity of hypoglycemia increases, the quality of life of patients decreases. Approximately 25% of patients with type 2 diabetes treated with insulin for more than five years experience severe hypoglycemia. Impaired awareness of hypoglycemia is the weakening of the ability to perceive warning signs during hypoglycemia. Impaired awareness of hypoglycemia is associated with a 6- to 9-fold increase in the risk of severe hypoglycemia. Recurrent hypoglycemia, defined as the occurrence of more than one hypoglycemic event, increases the risk of severe hypoglycemia, and this also reduces hypoglycemia awareness. Before implementing strategies to help increase hypoglycemia awareness in individuals with diabetes, it is important to identify individuals who are at risk for severe hypoglycemia or have decreased hypoglycemia awareness. The risk of severe hypoglycemia is highest in individuals who have had a severe hypoglycemic episode in the past or in patients with reduced awareness of hypoglycemia. Comprehensive interventions need to be developed to increase hypoglycemia awareness in diabetic patients. While structured and comprehensive hypoglycemia awareness training is limited even for individuals with type 1 diabetes in the literature, there is no training program specifically developed for type 2 diabetes. In line with this information, it is necessary to develop a structured training program for individuals with type 2 diabetes and reduced hypoglycemia awareness and evaluate its effectiveness. Therefore, the aim of this study is to examine the effect of the hypoglycemia prevention and awareness program (HypoPAP) on patient outcomes in individuals with type 2 diabetes with decreased hypoglycemia awareness. The study was planned as a randomized controlled study.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age and older
* Being able to communicate in Turkish
* Being diagnosed with type 2 diabetes
* Having used insulin for at least one year
* Having reduced hypoglycemia awareness
* Being willing to participate in the study
* Having and being able to use information technology products (telephone, computer).

Exclusion Criteria:

* Having visual, auditory, cognitive impairment
* Having a condition that prevents communication
* Not being able to use information technology products
* Having chronic renal failure, chronic vascular disease, chronic liver disease, cancer
* Pregnancy
* Endocrine and eating disorders
* Individuals who do not agree to participate in the study
* Do not meet the inclusion criteria will not be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
Hypoglycemic Confidence Scale | 1 month
  The Hypoglycemic Confidence Scale is a nine-item self-report scale developed by William Polonsky and colleagues in 2017 that examines the degree to which diabetic patients feel safe and comfortable about their ability to protect themselves from hypoglycemia-related problems. It was developed for use in adults with diabetes (Type 1 and Type 2 using insulin). The Hypoglycemic Confidence Scale focuses on three areas: 1. Self-confidence (e.g., confidence in recognizing and managing hypoglycemia before blood sugar drops too low) 2. Confidence in avoiding hypoglycemia at critical times (e.g., while driving, exercising, and sleeping) 3. An estimate of the confidence of the spouse/partner. The Hypoglycemic Confidence Scale items are scored between 1 and 4 (1; Not at all confident 2; Somewhat confident 3; Moderately confident 4; Very confident). The ninth scale item for diabetic individuals with a spouse was interpreted as: 1; Not at all confident 2; Somewhat confident 3; Moderately confident
Hypoglycemia Fear Scale | 1 month
  The Hypoglycemia Fear Survey-HFS, was used to determine the fear of hypoglycemia in diabetic individuals. This scale consists of two subgroups, behavior and anxiety, and a total of 33 items. The behavior subgroup of this scale consists of 15 items. In the behavior subgroup; diabetic individuals are asked questions about what they have done in their daily lives to prevent their blood glucose levels from falling in the last 6 months. The anxiety subgroup consists of 18 items, and individuals are asked how often they have worried about the items given due to low blood glucose levels in the last 6 months. The answers vary between; "0 points: never; 1 point: rarely; 2 points: sometimes; 3 points often; 4 points: always". A high score indicates a high fear of hypoglycemia.
Hypoglycemia Attitude and Behavior Scale | 1 month
  This scale was prepared for individuals with type 2 diabetes and consists of 14 items. It aims to measure hypoglycemia attitudes and behaviors of individuals with type 2 diabetes in three sub-dimensions: Avoidance (four items), confidence (five items) and anxiety (five items). Anxiety questions individuals' concerns about hypoglycemia. Avoidance questions the attitudes and behaviors adopted to avoid hypoglycemia. Confidence consists of questions aimed at determining the degree of comfort provided by not experiencing problems caused by hypoglycemia. The scale does not have a total score: While the avoidance and anxiety sub-dimensions are scored directly (1 = Strongly disagree, 5 = Strongly agree), the Confidence sub-dimension is scored inversely (1 = Strongly agree, 5 = Strongly disagree).
Hypoglycemia Awareness Questionnaire | 1 month
  The Hypoglycemia Awareness Questionnaire includes questions that evaluate the hypoglycemia awareness of the individuals participating in the study, how often they experience hypoglycemia, the symptoms they experience during hypoglycemia, and how they intervene when these symptoms occur. In the study, the responses of individuals to the question "Can you feel low blood sugar?" are evaluated. Individuals are required to select one of the following responses: "always," "usually," "sometimes," or "never." Patients who only respond "always" are considered to have normal symptomatic awareness of hypoglycemia; those who respond "usually" are defined as having reduced hypoglycemia awareness, and those who respond "sometimes and never" are defined as having no hypoglycemia awareness. The questionnaire is one of the most frequently used assessment questionnaires in the literature for hypoglycemia awareness .

CONTACTS AND LOCATIONS:
Overall Officials: Merve M Dervişoğlu, MSc, Principal Investigator — Dokuz Eylul University
Locations (1):
- Dokuz Eylül University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No